CLINICAL TRIAL: NCT04641455
Title: Use of Mucolytic Solution Before Upper Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Michal Štěpán, M.D., Principal investigator, Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DDC VN 10
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer; Gastroscopy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Espumisan; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A mucolytic solution (Experimental): mucolytic solution - 100 ml of water + 600 mg of N-acetylcysteine (3 tablets of 200 mg ACC long), 320 mg of simethicone (8 ml of Espumisan sir. 40 mg / ml)administered 20-30 minutes prior to upper endoscopy
  Interventions: Drug: Espumisan, N acetylcystein
- B mucolytic solution (Active Comparator): mucolytic solution-100 ml water + 400 mg N-acetylcysteine (2 tablets 200 mg ACC long), 20 mg simethicone (0.5 ml Espumisan sir. 40 mg / ml) administered 20-30 minutes prior to upper endoscopy
  Interventions: Drug: Espumisan, N acetylcystein
- C Water (Placebo Comparator): 100 ml of water 20-30 minutes prior to upper endoscopy
  Interventions: Drug: Water
- D No intervention (No Intervention): Upper endoscopy without neither mucolytic solution nor water prior to upper endoscopy.

INTERVENTIONS:
Drug: Espumisan, N acetylcystein — Administration of mucolytic solution before upper endoscopy (Espumisan 320 mg, ACC long 600 mg)
  Arms: A mucolytic solution
Drug: Espumisan, N acetylcystein — Administration of mucolytic solution before upper endoscopy (Espumisan 20 mg, ACC long 200 mg)
  Arms: B mucolytic solution
Drug: Water — Administration of water before upper endoscopy
  Arms: C Water

SUMMARY:
The study was designed to evaluate the effectiveness of the maximum dose of mucolytic solution used before upper endoscopy on the visibility of the gastric mucosa

DETAILED DESCRIPTION:
Residual gastric content containing mucus, bubbles, bile and food particles may limit visibility of gastric mucosa and therefore diagnostic yield of upper endoscopy, especially in cases of early neoplastic lesions. Data on benefit of peroral mucolytic solution administered before upper endoscopy are limited.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, signed informed consent, diagnostic gastroscopy

Exclusion Criteria:

* age < 18 years, interventional gastroscopy, known disease of the upper GI tract and/or history of surgery of GI tract, gastroscopy indicated of bleeding, dysphagia or ileus, liver cirrhosis, general anesthesia, allergy to mucolytic solution components, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Visibility score" evaluated by blinded performing endoscopist | through study completion, an average of 5 months
  Visibility score" (0-25 points) counted as the sum of visibility score in the esophagus (0-5), fundus (0-5), corpus (0-5) and atrum (0-5) of the stomach and in the duodenum (0-5).

SECONDARY OUTCOMES:
Visibility score" evaluated by two blinded endoscopists using 10 endoscopic images captured during endoscopy | through study completion, an average of 5 months
  "Visibility score" (0-25 points) counted as the sum of visibility score in the esophagus (0-5), fundus (0-5), corpus (0-5) and atrum (0-5) of the stomach and in the duodenum (0-5).

OTHER OUTCOMES:
Residual fluid in the stomach evaluated by blinded performing endoscopist | through study completion, an average of 5 months
  0-3 point scale
Duration of endoscopy | through study completion, an average of 5 months
  time between introduction and withdrawal of the endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michal Stepan, M.D., Principal Investigator — Digestive Diseases Center, Vítkovice Hospital
Locations (1):
- Digestive Diseases Center, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No